CLINICAL TRIAL: NCT02469155
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled, Multi-Center Study to Assess the Antipsychotic Efficacy of ITI-007 After 6 Weeks of Treatment in Patients With Schizophrenia
Brief Title: A Trial to Assess the Antipsychotic Efficacy of ITI-007 Over 6 Weeks of Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITI-007-302
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — lumateperone; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Lumateperone 14 mg (ITI-007 20 mg Tosylate) (Experimental): Lumateperone 14 mg (ITI-007 20 mg Tosylate) administered orally as formulated capsules once daily for 6 weeks
  Interventions: Drug: ITI-007
- Lumateperone 42 mg (ITI-007 60 mg Tosylate) (Experimental): Lumateperone 42 mg (ITI-007 60 mg Tosylate) administered orally as formulated capsules once daily for 6 weeks
  Interventions: Drug: ITI-007
- Placebo (Placebo Comparator): Placebo administered orally as visually-matched capsules once daily for 6 weeks
  Interventions: Drug: Placebo
- Risperidone (Active Comparator): Risperidone administered orally as visually-matched over-encapsulated tablet once daily for 6 weeks
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: ITI-007
  Arms: Lumateperone 14 mg (ITI-007 20 mg Tosylate); Lumateperone 42 mg (ITI-007 60 mg Tosylate)
Drug: Risperidone
  Arms: Risperidone
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study will evaluate the antipsychotic efficacy of ITI-007 in a randomized, double-blind, parallel-group, placebo- and active-controlled, multi-center study in patients diagnosed with schizophrenia having an acute exacerbation of psychosis.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects of any race, ages 18-60 inclusive, with a clinical diagnosis of schizophrenia
* experiencing an acute exacerbation of psychosis

Exclusion Criteria:

* any subject unable to provide informed consent
* any female subject who is pregnant or breast-feeding
* any subject judged to be medically inappropriate for study participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 696 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Vanover, Ph.D., Study Director — Intra-Cellular Therapies, Inc.
Locations (11):
- United States (11):
  - Clinical Site, Little Rock, Arkansas
  - Clinical Site, Springdale, Arkansas
  - Clinical Site, Culver City, California
  - Clinical Site, Lemon Grove, California
  - Clinical Site, Long Beach, California
  - Clinical Site, San Diego, California
  - Clinical Site, North Miami, Florida
  - Clinical Site, Berlin, New Jersey
  - Clinical Site, Marlton, New Jersey
  - Clinical Site, Austin, Texas
  - Clinical Site, Dallas, Texas

REFERENCES:
- [Derived] Citrome L, Durgam S, Edwards JB, Davis RE. Lumateperone for the Treatment of Schizophrenia: Number Needed to Treat, Number Needed to Harm, and Likelihood to Be Helped or Harmed. J Clin Psychiatry. 2023 Mar 6;84(2):22r14631. doi: 10.4088/JCP.22r14631. PMID 36883881

RESULTS

PARTICIPANT FLOW:
Groups:
- Lumateperone 14 mg (ITI-007 20 mg Tosylate): Lumateperone 14 mg (ITI-007 20 mg Tosylate) administered orally as formulated capsules once daily for 6 weeks
  ITI-007
- Lumateperone 42 mg (ITI-007 60 mg Tosylate): Lumateperone 42 mg (ITI-007 60 mg Tosylate) administered orally as formulated capsules once daily for 6 weeks
  ITI-007
- Placebo: Placebo administered orally as visually-matched capsules once daily for 6 weeks
  Placebo
- Risperidone: Risperidone administered orally as visually-matched over-encapsulated tablet once daily for 6 weeks
  Risperidone
Period: Overall Study
Arm/Group | Lumateperone 14 mg (ITI-007 20 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo | Risperidone
Started | 174 | 174 | 174 | 174
Completed | 113 | 128 | 133 | 105
Not Completed | 61 | 46 | 41 | 69
Not completed — Adverse Event | 6 | 0 | 1 | 10
Not completed — Lack of Efficacy | 13 | 10 | 10 | 8
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 5 | 2 | 7 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 34 | 30 | 20 | 37
Not completed — Other | 3 | 3 | 2 | 10
Not completed — Protocol Violation | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 4 subjects received an incorrect treatment compared to that which they were randomized. The numbers presented in Baseline Characteristics are as treated in each group except as noted.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lumateperone 14 mg (ITI-007 20 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo | Risperidone | Total
Number analyzed (Participants) | 172 | 172 | 178 | 173 | 695
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (9.99) | 41.9 (9.88) | 43.5 (9.90) | 42.4 (10.77) | 42.6 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 49 | 46 | 41 | 183
  Male | 125 | 123 | 132 | 132 | 512
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26 | 30 | 35 | 40 | 131
  Back or African American | 140 | 140 | 133 | 123 | 536
  Asian | 2 | 0 | 3 | 2 | 7
  Other | 4 | 2 | 7 | 8 | 21
Positive and Negative Syndrome Scale (PANSS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The PANSS is a 30-item scale used to measure symptoms of schizophrenia. The scale has 7 positive symptom items, 7 negative symptom items, and 16 general psychopathology symptom items. Each item is scored on a 7-point scale by the clinical rater based on a clinical interview with the patient, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms. Thus, the PANSS Total score minimum is 30 and the maximum is 210, with higher numbers indicating more severe symptoms.
  units on a scale | 88.7 (9.86) | 90.9 (10.26) | 90.0 (9.81) | 90.0 (9.60) | 89.9 (9.89)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS is a 30-item scale used to measure symptoms of schizophrenia. The scale has 7 positive symptom items, 7 negative symptom items, and 16 general psychopathology symptom items. Each item is scored on a 7-point scale by the clinical rater based on a clinical interview with the patient, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms. Thus, the PANSS Total score minimum is 30 and the maximum is 210, with higher numbers indicating more severe symptoms.
Time Frame: 6 weeks
Population: Analysis was conducted using the ITT analysis set, which includes all subjects who were randomized, received at least 1 dose of study medication, and had a valid baseline and at least 1 valid post-baseline PANSS measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lumateperone 14 mg (ITI-007 20 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo | Risperidone
Number analyzed (Participants) | 166 | 162 | 169 | 157
units on a scale | -15.0 (1.27) | -14.6 (1.23) | -15.1 (1.21) | -20.5 (1.33)
Statistical Analysis 1: Comparison: Lumateperone 14 mg (ITI-007 20 mg Tosylate) vs Placebo; Test type: Superiority; p = 0.972, Mixed Models for Repeated Measure; Least Squares Mean Difference = 0.1, 95% CI 2-sided [-3.39 to 3.51]
Statistical Analysis 2: Comparison: Lumateperone 42 mg (ITI-007 60 mg Tosylate) vs Placebo; Test type: Superiority; p = 0.789, Mixed Effects Model for Repeated Measure; Least Squares Mean Difference = 0.5, 95% CI 2-sided [-2.92 to 3.84]

2. Secondary Outcome: Change From Baseline to Week 6 in Clinical Global Impressions-Severity of Illness Scale
Description: The Clinical Global Impressions (CGI) Scale is a standardized assessment tool that the clinician can use to rate the severity of illness, change over time, and efficacy of medication, taking into account the subject's clinical condition and the severity of side effects. The CGI Scale consists of 3 global subscales, only one of which was used in the present study. The first subscale, Severity of Illness (CGI-S), assesses the clinician's impression of the subject's current illness state; it is often used both before and after treatment. Scores on the Severity of Illness subscale range from 1 = "not ill" at all to 7 = "among the most extremely ill."
Time Frame: 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From signing ICF until end of study procedures (~10 weeks), including 6 weeks of double blind treatment.
Description: 4 subjects received an incorrect treatment compared to that which they were randomized. The numbers presented are as treated in each group.
Arm/Group | Lumateperone 14 mg (ITI-007 20 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo | Risperidone
All-Cause Mortality (participants affected / at risk) | 0/172 | 0/172 | 0/178 | 1/173
Serious Adverse Events (participants affected / at risk) | 0/172 | 1/172 | 0/178 | 0/173
Other Adverse Events (participants affected / at risk) | 57/172 | 76/172 | 68/178 | 79/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lumateperone 14 mg (ITI-007 20 mg Tosylate) (N=172) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) (N=172) | Placebo (N=178) | Risperidone (N=173)
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 — Agitation (secondary to psychosis)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lumateperone 14 mg (ITI-007 20 mg Tosylate) (N=172) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) (N=172) | Placebo (N=178) | Risperidone (N=173)
Headache (Nervous system disorders) | 16 | 36 | 25 | 36
Somnolence (Nervous system disorders) | 19 | 31 | 11 | 30
Nausea (Gastrointestinal disorders) | 7 | 16 | 8 | 15
Constipation (Gastrointestinal disorders) | 10 | 12 | 17 | 7
Dyspepsia (Gastrointestinal disorders) | 6 | 9 | 10 | 3
Dry Mouth (Gastrointestinal disorders) | 4 | 9 | 0 | 7
Sedation (Nervous system disorders) | 11 | 7 | 5 | 14
Toothache (Gastrointestinal disorders) | 5 | 7 | 11 | 8
Weight Increased (Investigations) | 5 | 3 | 4 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes